CLINICAL TRIAL: NCT05605210
Title: Stimulation Sites and Fatigue Induced by Neuromuscular Electrical Stimulation in Healthy Individuals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marco Aurélio Vaz, PhD (Other)
Responsible Party: Sponsor-Investigator, Marco Aurélio Vaz, PhD, Principal Investigator, Federal University of Rio Grande do Sul
Organization: Federal University of Rio Grande do Sul (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 5.309.992
Record Dates: First submitted 2022-10-06; First posted 2022-11-04 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Fatigue
Keywords: Electrical stimulation; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- FN-NMES - 20 Hz (Experimental): This group will receive a NMES-induced fatigue protocol, which will be applied to the femoral nerve (FN) using a stimulation frequency of 20 Hz. For this, the participant will be positioned on the isokinetic dynamometer (Biodex Medical System, Shirley - NY, USA) with the knee in 90° of flexion (0°=total extension). The participant will be instructed to remain relaxed and to not perform active muscle contraction.
  Interventions: Device: Electric stimulation
- FN-NMES - 100 Hz (Experimental): This group will receive a NMES-induced fatigue protocol, which will be applied to the femoral nerve (FN) using a stimulation frequency of 100 Hz. For this, the participant will be positioned on the isokinetic dynamometer (Biodex Medical System, Shirley - NY, USA) with the knee in 90° of flexion (0°=total extension). The participant will be instructed to remain relaxed and to not perform active muscle contractions.
  Interventions: Device: Electric stimulation
- MP-NMES - 20 Hz (Experimental): This arm will receive a NMES-induced fatigue protocol, which will be applied to the motor point (MP) of the rectus femoris muscle using a stimulation frequency of 20 Hz. For this, the participant will be positioned on the isokinetic dynamometer (Biodex Medical System, Shirley - NY, USA) with the knee at 90° of flexion (0°=total extension). The participant will be instructed to remain relaxed and to not perform active muscle contractions.
  Interventions: Device: Electric stimulation
- MP-NMES - 100 Hz (Experimental): This arm will receive a NMES-induced fatigue protocol, which will be applied to the motor point (MP) of the rectus femoris muscle using a stimulation frequency of 100 Hz. For this, the participant will be positioned on the isokinetic dynamometer (Biodex Medical System, Shirley - NY, USA) with the knee at 90° of flexion (0°=total extension). The participant will be instructed to remain relaxed and to not perform active muscle contractions.
  Interventions: Device: Electric stimulation
- FNMP-NMES - 20 Hz (Experimental): This group will receive a NMES-induced fatigue protocol, which will be applied to the femoral nerve (FN) and to the motor point (MP) of the rectus femoris muscle using a stimulation frequency of 20 Hz. For this, the participant will be positioned on the isokinetic dynamometer (Biodex Medical System, Shirley - NY, USA) with the knee at 90° of flexion (0°=total extension). The participant will be instructed to remain relaxed and to not perform active muscle contractions.
  Interventions: Device: Electric stimulation
- FNMP-NMES - 100 Hz (Experimental): This group will receive a NMES-induced fatigue protocol, which will be applied to the femoral nerve (FN) and to the motor point (MP) of the rectus femoris muscle using a stimulation frequency of 100 Hz. For this, the participant will be positioned on the isokinetic dynamometer (Biodex Medical System, Shirley - NY, USA) with the knee at 90° of flexion (0°=total extension). The participant will be instructed to remain relaxed and to not perform active muscle contractions.
  Interventions: Device: Electric stimulation

INTERVENTIONS:
Device: Electric stimulation — Neuromuscular electrical stimulation will be applied at two sites to induce fatigue with stimulation frequency specified at the Arm/Group Descriptions. The electrical stimulation parameters to generate the fatigue protocol will be: biphasic pulsed current, pulse duration of 2 ms, and on:off times of 5:10s. The fatigue protocol will be applied with a current intensity sufficient to generate an evoked torque at a level of 20% of the MVIC, which will be maintained throughout the protocol. NMES will be maintained until reaching an intervention time of 20 minutes, generating 80 evoked contractions.

SUMMARY:
Neuromuscular electrical stimulation (NMES) is a tool used in training protocols and in clinical practice to prevent or attenuate atrophy and improve the ability to produce muscle strength in different populations. Although widely used, the effects of NMES can be limited by discomfort and early fatigue induced by electrical current. Previous studies have investigated alternatives to minimize muscle fatigue, reduce muscle discomfort and increase muscle performance. A measure adopted to reduce the NMES's deleterious effects is the choice of stimulation site. More specifically, muscle contractions can be evoked by applying electrical pulses to the trunk of peripheral nerves (nNMES) or terminal branches of the nerve at the muscle belly level (mNMES). There is evidence that the mNMES stimulates the more superficial motor units (MUs), while the deeper MUs of the muscle remain inactivated, or, to recruit them, an additional increase in current intensity and stimulation frequency may be required. On the other hand, in direct nerve stimulation (nNMES) both superficial and deep MUs are recruited regardless of NMES intensity. Based on these observations, a new application modality of NMES emerged, the intercalated nerve and muscle stimulation (iNMES). In this strategy, electrical pulses are intercalated or alternated between the mNMES and nNMES sites, intending to reduce the high frequencies at which the MUs are activated during NMES, recruiting both superficial and deep MUs, and reducing muscle fatigue during evoked contractions. Although iEENM is a promising strategy to potentiate the NMES effects, few studies have investigated the iNMES effects on neuromuscular fatigue, and the existing literature is solely focused on the analysis of the tibialis anterior muscle, limiting the findings' inferences for other muscles important for lower limb functionality (e.g., quadriceps femoris). Therefore, the objective of this study is to compare the effects of nNMES applied to the femoral nerve (FN-NMES), of mNMES applied to the rectus femoris' motor point (MP-NMES), and iNMES applied simultaneously to both sites (FNMP-NMES) on knee extensors' functional (muscle fatigue) and clinical (discomfort) parameters in healthy individuals, through a randomized clinical trial. Our study has three hypotheses. In our first hypothesis, muscle fatigue during an electrical stimulation protocol will be lower with the FNMP-NMES modality, followed by FN-NMES, and will be higher with MP-NMES. Thus, FNMP-NMES will present a smaller reduction in maximal voluntary isometric contractions (MVICs) immediately after the fatigue protocol, a smaller relative reduction between the final compared to the initial evoked torque, a greater number of contractions for the evoked torque to reduce 50% with respect to the initial torque during the NMES fatigue protocol, and a greater total work compared the FN-NMES and MP-NMES modalities. In our second hypothesis, low frequency (20 Hz) NMES will produce greater total work and less fatigability of the knee extensors (smaller reduction from pre to post MVIC, smaller percentage reduction at the final compared to the initial evoked torque, a greater number of contractions for the evoked torque to reduce 50% compared to the initial evoked torque, and greater total work) compared to a high stimulation frequency (100 Hz). Furthermore, the total work will be higher and the fatigability lower with FNMP-NMES, followed by FN-NMES, and finally MP-NMES, regardless of stimulation frequency. Finally, the third hypothesis is that discomfort will be less with FNMP-NMES, followed by FN-NMES, and finally MP-NMES, regardless of stimulation frequency.

DETAILED DESCRIPTION:
This project will be developed through one randomized clinical study, which will be designed to compare the effects of nNMES applied to the femoral nerve (NF-NMES), mNMES applied to the motor point (PM-NMES), and iEENM applied simultaneously at both sites (NFPM-NMES), using low (20Hz) and high (100 Hz) stimulation frequency, on knee extensors' fatigability and discomfort in healthy subjects. Therefore, this study is characterized by a quantitative approach with a randomized clinical cross-over design, blinded to evaluators and participants.

The sample will be characterized by convenience, and healthy men and women (self-declaration that they do not have diseases), aged between 18 and 40 years, will be recruited. To define the sample size, the G-Power software (version 3.1.3; University of Trier, Trier, Germany) was used, and a significance level was adopted for α = 0.05 and power (1-β) = 0.80, for all calculated variables. As the fatigability variable demonstrated the need for a larger sample (24 participants) to avoid errors and reach a minimum statistical power of 80%, the investigators will use the result of this variable for the present study. However, a previous study (DANTAS et al., 2015) reported the exclusion of 25% of individuals who were recruited for evaluation, for reasons related to NMES. Therefore, considering possible exclusions or even losses throughout the protocol, the investigators will recruit 30 participants throughout the study, 15 men and 15 women.

Assessments will be carried out on 6 different days for each participant. The duration of each evaluation will have an average time of 2 hours for the first evaluation day, and 1.5 hours for the other evaluation days. Additionally, women will be evaluated between the 4th and 22nd day of the menstrual cycle, a period in which there is a greater tolerance to NMES. On the first day, anamnesis will be carried out, explanations about the study will be provided and the participant will be familiarized with the assessment techniques and the assessment protocol. After this initial part, an interval of 10 minutes will be observed, and, then, the envelope will be opened containing which application protocol was randomized to be investigated, that is, tests using FN-NMES, MP-NMES, or FNMP-NMES, after which the following steps/tests will be applied:

1. Preparing participants for the tests;
2. Assessment of the supramaximal evoked twitch torque at rest;
3. Assessment of the maximum torque generated during maximal voluntary isometric contraction (MVIC) pre-fatigue;
4. Assessment of the supramaximal evoked twitch torque pre-fatigue;
5. Evaluation of the current intensity to generate a torque at 20% of the MVIC;
6. Application of the NMES-evoked fatigue protocol;
7. Assessment of discomfort during the fatigue protocol;
8. Evaluation of the maximum torque generated during the MVIC after fatigue;
9. Assessment of the supramaximal evoked twitch torque after the fatigue protocol. This study will adopt an intention-to-treat approach. Therefore, the individual who does not attend the scheduled evaluation will be rescheduled for a new evaluation, allowing the individual to carry out all scheduled evaluations. If the subject chooses to withdraw from participating in the research project, the data collected until the end of his/her participation in the study will be used for analysis. Thus, a flowchart will be used to indicate the abandonment of subjects during all phases of the study, if it does occur. In addition, the flowchart will record how individuals will be included/excluded in the different phases of the study. The statistical procedures will be performed in the SPSS 21.0 program for Windows, and the data tabulation in the Excel 2016 program. The distribution of variables will be presented as mean and standard deviation. The Shapiro-Wilk test will be used to analyze the normality of the data distribution. To compare the fatigability between NMES modalities, ANOVA will be used for repeated measures of two intramodality factors (NMES frequencies and pre/post-NMES protocol time) and an intermodality factor (gender). To compare discomfort between NMES modalities, ANOVA will be used for repeated measures of two intramodality factors (NMES frequencies and NMES site) and an intermodality factor (gender). If there is an interaction between factors, a one-way ANOVA for repeated measures will be used to see if there are differences between the modalities, and, to locate the differences, the Bonferroni post hoc test will be used. In addition, the Cohen's "d" effect size will be calculated, which will be categorized as trivial (<0.20), small (0.20-0.49), moderate (0.50-0.79), large (0.80 to 1.29), and very large. (>1.30) (ROSENTHAL, 1996).

ELIGIBILITY:
Inclusion Criteria:

Healthy individuals:

1. young people of both sexes
2. age between 18 and 40 years
3. body mass index between 20 and 25 kg/m2
4. and normal knee range of motion
5. with no complaints of pain or presence of pathology in the dominant lower limb. -

Exclusion Criteria:

Individuals with:

1. any contraindication to maximal exercise
2. having been treated with NMES in the last 3 months in the lower limb
3. not tolerate electrical stimulation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Level of physical activity | The assessment will be performed before the introduction of the intervention.
  The level of physical activity (PA) of each subject will be assessed by the International Physical Activity Questionnaire (IPAQ).The scores will be assessed by calculating the metabolic equivalents (MET) for each activity level. Walking score will be achieved by the multiplication of 3.3 METs with the total walking duration in minutes in a week. Moderate physical activity scores will be achieved by the multiplication of 4.0 METs with the total moderate physical activity duration in minutes in a week. Vigorous physical activity scores will be achieved by the multiplication of 8.0 METs with the total vigorous physical activity duration in minutes in a week. Total physical activity MET-minutes/week will be obtained through sum of walking, moderate and vigorous MET minutes/week scores. Categorical Score will be classified into three levels of physical activity: low, moderate and high.
Thickness of the subcutaneous fat layer on the motor point and femoral nerve | The assessment will be performed pre-intervention, that is, before each NMES protocol
  Corresponds to the amount of subcutaneous adipose tissue and will be evaluated by ultrasonography
Maximum voluntary isometric contraction of the knee extensors | The assessment will be performed pre-intervention, that is, before each NMES protocol
  Knee extensor maximal voluntary isometric contraction (MVIC) is an expression of the muscular strength, and will be evaluated by dynamometry.
Current intensity required to evoke knee extensors' submaximal torque (20% MVIC) | The assessment will be performed pre-intervention, that is, before each NMES protocol
  The amount or amplitude of electrical current (in milliamperes - mA) required to achieve a specific force (20% MVIC), and will be evaluated from the electrical stimulation device.
Change from rest Evoked torque by supramaximal twitch at pre-intervention and immediately after the intervention | This evaluation will be carried out at rest, pre-intervention and immediately after the intervention
  Simple biphasic rectangular electrical pulses will be applied at a frequency of 1 Hz at a current intensity sufficient to generate a visible contraction of the knee extensors. From the identification of this motor threshold, the current intensity will be gradually increased until no subsequent increase in the evoked twitch torque is observed. Then, the current intensity will be increased by 10% in order to guarantee that the torque evoked by the twitch is supramaximal. The torque (Nm) evoked during the twitch will be determined by the torque produced by three supramaximal stimuli.
Muscle Fatigue Index | During 5 sec minutes before and after of electrical stimulation protocol
  Characterized by the maximal voluntary isometric contraction decrease after the fatigue protocol, it will be evaluated by dynamometry.
Fatigue Index from Evoked Torque | During 20 minutes of electrical stimulation
  Characterized by the decrease of the evoked torque during the fatigue protocol, the fatigue index from the evoked torque will be evaluated by dynamometry, and obtained by the analysis of evoked torque curves
Reduction of the torque evoked until reaching 50% of the torque evoked by the first contraction | During 20 minutes of electrical stimulation
  It will be obtained from the analysis of the evoked contractions' torque-time curves. The torque evoked by each contraction will be normalized by the torque evoked by the first contraction (which will correspond to 100%). The number of contractions until the relative evoked torque to undergo a 50% reduction in relation to the evoked torque of the initial contraction will be used for analysis.
Total work generated during the fatigue protocol | During 20 minutes of electrical stimulation
  The torque-time integral of the evoked torque curves during the fatigue protocol will be evaluated and correspond to the mechanical work of each evoked contraction. The sum of the torque curve integral of all evoked contractions during the fatigue protocol will be calculated to determine the total work evoked by each current during the fatigue protocol.
Discomfort level generated by electrical stimulation during the fatigue protocol | During 20 minutes of electrical stimulation
  Discomfort will be measured with a Visual Analogue Scale (0-100mm), where 0 and 100 mm correspond to no discomfort and worst perceived discomfort, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Vaz, PhD, Principal Investigator — Federal University of Rio Grande do Sul; Marco A Vaz, PhD, Study Chair — Federal University of Rio Grande do Sul; Marco A Vaz, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Exercise Research Laboratory, School of Physical Education, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil